CLINICAL TRIAL: NCT03086642
Title: Study of Talimogene Laherparepvec Administered Endoscopically for the Treatment of Locally Advanced or Metastatic Pancreas Cancer Refractory to at Least One Chemotherapy Regimen
Brief Title: Study of Talimogene Laherparepvec (T-VEC) in Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karie D. Runcie, MD (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Karie D. Runcie, MD, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAQ9966; 1R01FD006108-01 (FDA)
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Cancer
Keywords: locally advanced pancreatic cancer; locally advanced pancreas cancer; metastatic pancreatic cancer; metastatic pancreas cancer; refractory; refractory pancreatic cancer; refractory pancreas cancer; T-Vec; T Vec
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- T-Vec (Experimental): All enrolled patients will receive a test dose of talimogene laherparepvec (10^6 plaque forming units (PFU)/ml) on day 1, followed by treatment doses at escalating concentrations weeks 4, 7, and 10. A biopsy will be obtained during each scheduled endoscopy prior to talimogene laherparepvec injection.
  Interventions: Drug: Talimogene laherparepvec

INTERVENTIONS:
Drug: Talimogene laherparepvec — T-Vec will be administered by intratumoral injection into pancreatic tumors accessible endoscopically with ultrasound guidance (at least one pancreatic lesion must be injected during each treatment).
  On day 1 of week 1 the first dose of talimogene laherparepvec will be up to 4.0 mL of 10^6 PFU/mL. The second injection up to 4.0 mL of 10^6, 10^7, or 10^8 PFU/mL should be administered no sooner than day 1 of week 4 but should not be delayed more than 7 days after the scheduled time point. The maximum volume of T-Vec administered at any one time is 4.0 mL for any individual lesion.
  Other Names: T-Vec; T Vec

SUMMARY:
The purpose of this study is to find out which doses of talimogene laherparepvec (T-Vec) can be given safely to participants with pancreatic cancer that is either too big to be taken out by surgery or has spread to other parts of the body. The study will also see if T-Vec can cause tumor shrinkage or prevent its growth.

The primary objective is to determine the rate of dose limiting toxicity at tested doses of talimogene laherparepvec administered endoscopically to pancreatic tumors, and to identify a maximum tolerated dose (MTD).

Secondary exploratory efficacy endpoints include change in longest diameter in the injected lesion(s), overall response rate (ORR) per RECIST v1.1 and modified immune-related response criteria (mirRC as defined in section 11), progression free survival (PFS) and overall survival (OS) at 6, 12, and 24 months.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDA) is an area of great unmet need. PDA accounts for 90% of pancreatic tumors in 2016. The standard of care for pancreas cancer is cytotoxic chemotherapy, but this is not particularly effective with best response rates reported of 20-30% and no significant long-term 5-year survival for patients who are not surgical candidates. Talimogene laherparepvec (previously known as OncoVEXGM-CSF) is an intratumorally delivered oncolytic immunotherapy comprised of an immune-enhanced herpes simplex virus type-1 (HSV-1) that selectively replicates in solid tumors. Talimogene laherparepvec was the first oncolytic viral therapy to be approved by the Federal Drug Administration (FDA) for the treatment of cancer, specifically melanoma. There is the potential that talimogene laherparepvec could exert a systemic effect mitigating the potential of PDA to metastasize.

This is a phase 1 dose escalation study to evaluate the safety of talimogene laherparepvec in PDA. To find out which doses are safe, all participants enrolled in this study will receive up to 4 injections of T-Vec. At least two doses will be evaluated in this study, depending on how many side effects are seen at each dose. Participants will not be able to pick the dose, as this will be determined based on the study experience with participants enrolled previously.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have pathologically confirmed, locally advanced or metastatic pancreatic adenocarcinoma deemed surgically unresectable by a surgeon with expertise in pancreatic cancer
2. Disease must be refractory to or intolerant of at least first-line chemotherapy which contains 5-fluorouracil or gemcitabine
3. The primary lesion must be accessible for endoscopic biopsy and injection as evaluated by a gastroenterologist at NewYork Presbyterian -Columbia. Further, the patient must be deemed able to tolerate repeated endoscopy procedures by an anesthesiologist and/or gastroenterologist at NewYork Presbyterian-Columbia
4. Age 18 years or older
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
6. Radiologically measurable injectable disease in the pancreas or surgical bed from prior ≥1cm, as defined by RECIST v1.1
7. Ability to understand and the willingness to sign a written informed consent document
8. Females of child-bearing potential (defined as a sexually mature woman who (1) has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or (2) has not been naturally postmenopausal for at least 24 consecutive months [i.e., has had menses at any time during the preceding 24 consecutive months]) must:

   i. Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis), or agree to use, and be able to comply with, effective contraception (</=1% failure rate annually) without interruption, 28 days prior to starting therapy (including dose interruptions), and while on study medication or for a period of 30 days following treatment completion. [Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].

   ii. Have a negative urine or serum pregnancy test within 72 hours prior to enrollment. If urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.This applies even if the subject practices true abstinence from heterosexual contact.
9. Male subjects must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 30 days following treatment discontinuation, even if he has undergone a successful vasectomy.
10. Adequate organ and marrow function as defined below without need for hematopoietic growth factor or transfusion support:

    * Hemoglobin ≥8.0g/dl
    * Platelets ≥75,000/microliter (mcL)
    * Absolute neutrophil count (ANC) ≥1500/mm3 (1.5x109/L)
    * Total bilirubin ≤1.5 x institutional upper limit of normal (ULN) or Direct bilirubin ≤ ULN with total bilirubin >1.5 x ULN
    * Aspartate aminotransferase (AST) (SGOT)/alanine transaminase (ALT) (SGPT) ≤1.5 x ULN
    * INR and aPTT ≤ 1.5 x ULN Unless the patient is on therapeutic anticoagulation in which case the international normalized ratio (INR) and activated partial thromboplastin time (aPTT) must be within the therapeutic range of intended use of anti-coagulants
    * Serum creatinine ≤1.5 x ULN or 24 hour creatinine clearance ≥60 mL/min/1.73 m2 by Cockcroft-Gault
    * Lipase ≤3 x ULN

Exclusion Criteria:

1. Cystic pancreatic cancer. Microcystic disease may be eligible
2. Patients with pancreatic metastases deemed likely to limit the patient's ability to participate in the study for the complete duration (ie. >3 months), including but not limited to:

   a. Presence of central nervous system (CNS) metastasis including brain metastasis or compromise resulting from extrinsic disease in the bone or dura b. Presence of more than 5 liver metastases or one liver metastasis measuring more than 3cm c. Oxygen requirement attributable to pleural effusion or other malignant process d. Symptomatic ascites or radiographic evidence of more than trace ascites
3. History of other malignancy within the past 3 years with the following exceptions:

   1. malignancy treated with curative intent and with no known active disease present and has not received chemotherapy for >3 years before randomization and felt to be at low risk for recurrence by the treating physician
   2. adequately treated non-melanoma skin cancer without evidence of disease at the time of randomization • adequately treated cervical carcinoma in situ without evidence of disease at the time of randomization
   3. adequately treated breast ductal carcinoma in situ without evidence of disease at the time of randomization • prostatic intraepithelial neoplasia without evidence of prostate cancer at the time of randomization
   4. adequately treated superficial or in situ carcinoma of the bladder without evidence of disease at the time of randomization
4. Pancreatitis that is active or within the preceding 3 months which in the judgment of the endoscopist would make tumor injection likely to trigger severe recurrent pancreatitis.
5. Prior chemotherapy or radiotherapy within 14 days prior to first dose of therapy or has not recovered to CTCAE grade 1 or better from adverse event at time of enrollment due to cancer therapy administered more than 28 days prior to enrollment. or prior biological cancer therapy, targeted therapy, or major surgery within 28 days prior to first dose of therapy or unresolved grade 2 or greater toxicity from prior treatment, including chemotherapy, hormonal therapy, or radiotherapy, at the time of study enrollment. The following ongoing treatments are permitted:

   1. Hormone-replacement therapy or oral contraceptives
   2. Hormone therapy for primary prevention of breast cancer

5. Patients may not receive Coumadin while on study. Patients may receive low molecular weight heparin or novel oral anticoagulants (eg. dabigatran, apixaban, rivaroxaban) provided that the dose is held 1-2 days before injections are given and biopsies are performed per the protocol. Anti-platelet agents and herbal substances are allowed at the discretion of the treating endoscopist.

6. Radiation to the abdominal area within 28 days of first dose of therapy or prior radiotherapy in which the field does not overlap the injection sites or non-immunosuppressive targeted therapy within 14 days prior to enrollment or has not recovered to CTCAE grade 1 or better from adverse event due to cancer therapy administered more than 14 days prior to enrollment. .

7. The patient has not recovered to CTCAE grade 1 or better from adverse event at time of enrollment due to cancer therapy administered more than 28 days prior to enrollment

8. Prior biological cancer therapy, targeted therapy, or major surgery within 28 days prior to first dose of therapy or major surgery within 28 days prior to enrollment or has not recovered to CTCAE grade 1 or better from adverse event due to cancer therapy administered more than 28 days prior to enrollment. Adjuvant hormonal therapy is allowed..

9. Unresolved grade 2 or greater toxicity from most recent treatment, including chemotherapy, hormonal therapy, or radiotherapy, at the time of study enrollment.

10. The following ongoing treatments are permitted:

1. Hormone-replacement therapy or oral contraceptives
2. Hormone therapy for primary prevention of breast cancer

   11. Patients may not receive Coumadin while on study. Patients may receive low molecular weight heparin or novel oral anticoagulants (eg. dabigatran, apixiban, rivaroxaban) provided that the dose is held 1-2 days before injections are given and biopsies are performed per the protocol. Anti-platelet agents and herbal substances are allowed at the discretion of the treating endoscopist.

   12. Active herpetic skin lesions or prior complications of herpetic infection (e.g., herpetic keratitis or encephalitis) or requires intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (e.g., acyclovir), other than intermittent topical use.

   13. Previous treatment with talimogene laherparepvec or any other oncolytic virus

   14. Prior therapy with tumor vaccine

   15. Received live vaccine within 28 days of tumor enrollment

   16. Currently receiving treatment with another investigational device or drug study, or < 28 days since ending treatment with another investigational device or drug study(s). Other investigational procedures while participating in this study are excluded

   17. Known to have acute or chronic active hepatitis B infection, hepatitis C infection, or known to have human immunodeficiency virus (HIV) infection.

   18. Subject has known sensitivity to talimogene laherparepvec or any of its components to be administered during dosing.

   19. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection including Tuberculosis (TB) and C. difficile, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. This includes known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease

   20. Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia

   21. Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study

   22. Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during study treatment and through 3 months after the last dose of talimogene laherparepvec. (Note: Women not of childbearing potential are defined as: Any female who is post-menopausal [age > 55 years with cessation of menses for 12 or more months or less than 55 years but not spontaneous menses for at least 2 years or less than 55 years and spontaneous menses within the past 1 year, but currently amenorrheic (eg, spontaneous or secondary to hysterectomy), and with postmenopausal gonadotropin levels (luteinizing hormone and follicle-stimulating hormone levels > 40 IU/L) or postmenopausal estradiol levels (< 5 ng/dL) or according to the definition of "postmenopausal range" for the laboratory involved] or who have had a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy).

   23. Sexually active subjects and their partners unwilling to use male or female latex condom to avoid potential viral transmission during sexual contact while on treatment and within 30 days after treatment with talimogene laherparepvec.

   24. Nursing patients are not allowed on the study and women must commit to no lactation during the course of the study.

   25. Subject who is unwilling to minimize exposure with his/her blood or other body fluids to individuals who are at higher risks for HSV-1 induced complications such as immunosuppressed individuals, individuals known to have HIV infection, pregnant women, or children under the age of 1 year, during talimogene laherparepvec treatment and through 30 days after the last dose of talimogene laherparepvec.

   Immunotherapy-Related Exclusion Criteria:

   26. History or evidence of active autoimmune disease that requires systemic treatment (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment for patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation.
   * The use of inhaled or oral corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.

     27. Received live vaccine within 28 days prior to enrollment.

     28. Evidence of clinically significant immunosuppression such as the following:
   * Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease
   * HIV positive
   * Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 2 months prior to enrollment
   * Concurrent opportunistic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 36-48 months
  To determine the highest dose of study treatment that does not cause unacceptable side effects.

SECONDARY OUTCOMES:
Change in size of injected lesion(s) | baseline, 11 weeks
  To make an exploratory assessment of activity of talimogene laherparepvec in pancreatic cancer, as measured by change in size of the injected lesion(s)
Overall response rate (ORR) | Up to 24 months
  The percentage of patients whose cancer shrinks or disappears after treatment.
Progression-free survival (PFS) | Up to 24 months
  The length of time during and after the study treatment of cancer, that a patient lives with the disease but it does not get worse.
Overall survival (OS) | Up to 24 months
  The length of time from either the date of diagnosis or the start of study treatment for cancer, that patients diagnosed with the disease are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Karie Runcie, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Runcie K, Bracero Y, Samouha A, Manji G, Remotti HE, Gonda TA, Saenger Y. Phase I study of intratumoral injection of talimogene laherparepvec for the treatment of advanced pancreatic cancer. Oncologist. 2025 Jan 17;30(1):oyae200. doi: 10.1093/oncolo/oyae200. PMID 39673447
- See also: Cancer Center's clinical trials online search tool — http://www.hiccc.columbia.edu/ct/